CLINICAL TRIAL: NCT05252442
Title: An Assessment of a Relationship Between the Exposure to COVID-19 Vaccines and Risk of Thrombotic Thrombocytopenia Syndrome ATTEST Study (Association of the Risk for Thrombotic Thrombocytopenia Syndrome and Exposure To COVID-19 Vaccines)
Brief Title: Association of the Risk for Thrombotic Thrombocytopenia Syndrome and Exposure To COVID-19 Vaccines
Acronym: ATTEST
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8111R00010
Record Dates: First submitted 2022-01-24; First posted 2022-02-23 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-COVID-19
  Interventions: Other: Pre-COVID-19
- COVID-19
  Interventions: Other: COVID-19
- COVID-19 vaccination roll-out
  Interventions: Other: COVID-19 vaccination roll-out

INTERVENTIONS:
Other: Pre-COVID-19 — Pre-COVID-19 period
  Groups: Pre-COVID-19
Other: COVID-19 — COVID-19 period
  Groups: COVID-19
Other: COVID-19 vaccination roll-out — COVID-19 vaccination roll-out period
  Groups: COVID-19 vaccination roll-out

SUMMARY:
Background/Rationale: A very rare syndrome of thrombosis associated with low platelets has been reported in a few cases of recent exposure to COVID-19 vaccine. This thrombotic thrombocytopenia syndrome seems to be affecting patients of all ages and both genders; at present there is no clear signal of risk factors.

Objectives: To evaluate an association between COVID-19 vaccine exposure and thromboembolic events occurring with thrombocytopenia (thrombotic thrombocytopenia syndrome; TTS).

Study design: Two primary study designs will be considered, a case control study and a self-controlled case series (SCCS). A cohort analysis will be considered, in addition or as an alternative to either of the primary study designs, pending feasibility assessment of the follow-up time.

Data Source(s): Data for the study will be accessed through the NHS Digital Trusted Research Environment (TRE), providing national data coverage. Primary care data will be linked with vaccination, hospitalization, COVID-19 test results, mortality data. Initial exploratory analyses will be conducted using the Oxford-Royal College of General Practitioners sentinel network; ORCHID network database (N>15million).

Subjects of interest are patients who have received a COVID-19 vaccine. However, investigators will require access to data from all subjects in the databases.

Statistical Analysis: The study period will start on December 02, 2020, when the COVID-19 vaccine was first approved in the UK and will end at the end of data availability.

For the case-control design, all cases of TTS will be matched with control using risk-set matching. A case or matched control will be considered exposed if a COVID-19 vaccination will be within risk interval prior to the diagnosis date of the matched case.

For the SCCS, estimates of relative incidence (RI), in all risk intervals will be reported.

For the retrospective cohort design, the incidence of TTS after receiving COVID-19 vaccine will be estimated and investigators will compare this incidence with that occurring in an unvaccinated comparator group about levels of infection across the whole population.

Variables: Demographic, socioeconomic descriptors, clinical diagnosis, vaccines, potential confounders, thrombotic phenomena, COVID-19 infection, and other characteristics as applicable.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 12 months medical history prior to the start of the study period

Exclusion Criteria:

* Less than 12 moths medical history prior to the start of the study period

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 vaccinated English population with in one study historic and concurrent controls; and in the other a self-controlled case series.
Sampling Method: Non-Probability Sample
Enrollment: 7641136 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
thrombotic thrombocytopenia syndrome; TTS | 9 months
  This is to complete studies in NHS Digital and ORCHID data

CONTACTS AND LOCATIONS:
Locations (1):
- Research site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D8111R00010_Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111R00010&attachmentIdentifier=ac687de7-8521-42f5-b573-ad54daed8ddd&fileName=D8111R00010_Redacted_CSR_Synopsis.pdf&versionIdentifier=